CLINICAL TRIAL: NCT05176704
Title: Development and Validation of a Novel Functional Eye-Tracking Software Application for Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Innodem Neurosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ETNA-AD
Record Dates: First submitted 2021-12-03; First posted 2022-01-04 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Eye Movement Biomarkers; eye-tracking
MeSH Terms: conditions — Alzheimer Disease | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- CDR = 0.5: 50 Alzheimer's Disease (AD) patients including predominant AD with mixed vascular and MCI due to AD based on their CDR score. Questionable/very mild dementia (CDR = 0.5)
  Interventions: Device: Eye-Tracking
- CDR = 1: 50 Alzheimer's Disease (AD) patients including predominant AD with mixed vascular and MCI due to AD based on their CDR score. Mild dementia/MCI (CDR = 1)
  Interventions: Device: Eye-Tracking
- CDR = 2: 50 Alzheimer's Disease (AD) patients including predominant AD with mixed vascular and MCI due to AD based on their CDR score. Moderate dementia (CDR = 2)
  Interventions: Device: Eye-Tracking
- CDR = 3: 50 Alzheimer's Disease (AD) patients including predominant AD with mixed vascular and MCI due to AD based on their CDR score. Severe dementia (CDR = 3)
  Interventions: Device: Eye-Tracking
- Healthy Control: 50 Participant with no evidence or history of significant neurodegenerative disorder affecting brain function.
  Interventions: Device: Eye-Tracking

INTERVENTIONS:
Device: Eye-Tracking — Eye-tracking technology and algorithms used to successfully capture and track eye movements using an electronic tablet and the embedded camera of the device.

SUMMARY:
This study aims to develop and validate a sensitive and non-invasive eye-tracking software application.

This study will obtain participant responses to brief cognitive tests designed to evaluate several key functions known to be affected by Alzheimer's Disease and non-invasive eye movement measurements in response to visually presented stimuli during specifically designed eye-tracking tests. The study data will be used to develop machine learning algorithms and validate a software application intended to track the progressive component of Alzheimer's Disease and associated cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

  1. Able to provide informed consent
  2. Aged 18 years or older at the time of enrollment
  3. Able to read in either French or English
  4. Visual acuity of 20/100 in at least one eye (corrective glasses, contact lenses, surgery etc. are permitted)
* For patients only:

  1. Confirmed diagnosis of AD based on the NIAAA diagnostic criteria of probable AD
  2. Having undergone a full neuropsychological evaluation within the last 6 months or having a planned full neuropsychological evaluation within the next 6 months.
  3. AD diagnoses supported by FDG-PET scan or amyloid biomarkers (CSF or amyloid PET)

Exclusion Criteria:

* For AD participants:

  1. Diagnosed with one of the following dementia subtypes: Fronto-temporal dementia, Lewy-body dementia, or Creutzfeldt-Jakob disease.
  2. Incapacity to provide informed consent or inability to adequately understand the task instructions.
* For all participants:

  1. Evidence or medical history of psychiatric issues, which are known to also affect movements and oculomotor control.
  2. Presence of comorbid neurological conditions to avoid eye movement anomaly confounds (strabismus, cranial nerve palsy, stroke-causing hemianopsia).
  3. Diagnosis of macular edema or other pre-existing ocular conditions (e.g., glaucoma, cataracts) that would prevent from performing the eye movement assessments.
  4. Unstable medication use: recent (less than one month from enrollment) start of, change of dose, or irregular use of, new prescription drugs known to have an effect on ocular motor visual function, such as benzodiazepines, antipsychotics and anticonvulsants. Occasional use of benzodiazepines for medical procedures is permitted, at the investigator's discretion, but should not occur within a short time period of an eye movement assessment.
  5. Diagnosed with an active substance use disorder.
  6. History of stroke.
  7. Recent traumatic brain injury (within the last 6 months).
* For healthy controls only:

  1. Evidence or history of significant neurodegenerative disorder affecting brain function (e.g., MS, PD, ALS, Non-AD Dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this study, we will recruit 250 participants. 200 will be AD patients (including predominant AD with mixed vascular and MCI due to AD), who will subsequently be divided into 4 sub-groups of 50 based on their CDR score (questionable/very mild dementia (CDR = 0.5), mild dementia/MCI (CDR = 1), moderate dementia (CDR = 2), and severe dementia (CDR = 3)), and 50 will be healthy cognitively intact age-matched control participants.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating (CDR) score, one time, at the day of enrollment. | Baseline
  The Clinical Dementia Rating (CDR) is a global rating scale for staging patients diagnosed with Alzheimer disease and other dementias and monitoring changes in the level of there disabilities over time. The CDR scale is a 0-3 point numeric scale (0.5 unit increments) derived from clinician rating of cognition and daily function in the domains of memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care.

SECONDARY OUTCOMES:
The Montreal Cognitive Assessment (MoCA) score, one time, at the day of enrollment. | Baseline
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment and Alzheimer's disease. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.
The Mini-Mental State Exam (MMSE) score, one time, at the day of enrollment. | Baseline
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly, it includes tests of orientation, attention, memory, language and visual-spatial skills. It consists of a series of questions and tests that can be used by clinicians to help diagnose dementia and to help assess its progression and severity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Douglas Research Centre, Montreal, Quebec, Canada